CLINICAL TRIAL: NCT06409650
Title: A Phase II, Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Safety and Efficacy of KX-826 Tincture for Topical Use in Chinese Adult Female Patients With Androgenetic Alopecia (AGA)
Brief Title: To Evaluate Safety and Efficacy of KX-826 in Chinese Female Subjects With Androgenetic Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Koshine Biomedica, Inc. (Industry)
Responsible Party: Sponsor
Organization: Suzhou Kintor Pharmaceutical Inc, (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KX0826-CN-1004
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Alopecia
Keywords: Androgenetic Alopecia; Hair loss; Female pattern hair loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A (Experimental): KX-826 2.5mg QD
  Interventions: Drug: KX-826 dosed at 2.5mg
- Arm B (Experimental): KX-826 2.5mg BID
  Interventions: Drug: KX-826 dosed at 2.5mg
- Arm C (Experimental): KX-826 5mg QD
  Interventions: Drug: KX-826 dosed at 5 mg
- Arm D (Experimental): KX-826 5mg BID
  Interventions: Drug: KX-826 dosed at 5 mg
- Arm E (Placebo Comparator): Matching placebo QD
  Interventions: Drug: Matching placebo to KX-826
- Arm F (Placebo Comparator): Matching placebo BID
  Interventions: Drug: Matching placebo to KX-826

INTERVENTIONS:
Drug: KX-826 dosed at 2.5mg — 2.5mg of the investigational drug to be applied topically to scalp once daily for 24 weeks
  Arms: Arm A
Drug: KX-826 dosed at 2.5mg — 2.5mg of the investigational drug to be applied topically to scalp twice daily for 24 weeks
  Arms: Arm B
Drug: KX-826 dosed at 5 mg — 5mg of the investigational drug to be applied topically to scalp once daily for 24 weeks
  Arms: Arm C
Drug: KX-826 dosed at 5 mg — 5mg of the investigational drug to be applied topically to scalp twice daily for 24 weeks
  Arms: Arm D
Drug: Matching placebo to KX-826 — Placebo applied topically to scalp once daily for 24 weeks
  Arms: Arm E
Drug: Matching placebo to KX-826 — Placebo applied topically to scalp twice daily for 24 weeks
  Arms: Arm F

SUMMARY:
This was a multi-center, randomized, double-blind, placebo-controlled Phase II clinical study of KX-826 Tincture in Chinese adult female subjects with AGA.

DETAILED DESCRIPTION:
KX-826 is a new investigational androgen receptor (AR) antagonist for the treatment of female pattern hair loss (androgenetic alopecia). A total of 160 female subjects were randomized to one of four cohorts: 2.5 mg QD, 2.5 mg BID, 5 mg QD, 5mg BID of KX-826 or placebo (BID or QD) for 24 weeks. The primary endpoint of the study is to assess the changes from baseline in non-vellus TAHC （Target Area Hair Counts）at Week 24 in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria may be included in this study:

  1. Agree to follow the study treatment regimen and visit plan, voluntarily enroll in the study and sign the ICF in writing;
  2. Female, ≥ 18 years old;
  3. Clinically diagnosed as androgenetic alopecia;
  4. Alopecia severity was Ggraded D3-D6 according toon Savin scale;
  5. Willing to maintain the same hair style, color and length at each follow-up visit;
  6. Have no pregnancy plan and agree to take highly effective contraceptives throughout the study and within 3 months after the last dose. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study drug.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from the study:

  1. Medical/surgical history of any uncontrolled serious clinical system diseases, which may affect the safety and efficacy evaluation of the study drug, such as circulatory system, nervous system, hematological system, digestive system (e.g., inflammatory bowel disease), immune system, psychiatric disorders, etc.;
  2. Known hair loss disorders other than AGA, such as alopecia areata or diffuse alopecia areata, syphilitic alopecia, cicatricial alopecia, malnutrition, alopecia due to chemotherapy/radiotherapy;
  3. Scalp skin diseases that affect the efficacy evaluation, scalp trauma, or other scalp skin lesions requiring topical drug therapy, such as fungal or bacterial infection, severe seborrheic dermatitis, scalp psoriasis, contact dermatitis, severe folliculitis and scalp atrophy;
  4. Concomitant diseases that affect hair growth, such as connective tissue disease, inflammatory bowel disease, moderate to severe anemia and significant short-term weight loss;
  5. History of hair transplantation or requiring long-term wearing of a wig and hair adhesive during the study treatment;
  6. Have used topical drugs for hair loss sites (including corticosteroids, estrogens, etc.) that may affect the efficacy evaluation for ≥ 2 consecutive weeks within 3 months prior to screening;
  7. Have used androgen replacement therapy, immunosuppressants and other drugs that may affect the efficacy evaluation within 3 months prior to screening;
  8. Have used minoxidil within 6 months prior to screening;
  9. Have used spironolactone or cyproterone within 6 months prior to screening;
  10. Have received autologous platelet-rich plasma therapy for AGA within 12 months prior to screening;
  11. Have received chemotherapy and cytotoxic agents within 12 months prior to screening or have received scalp radiation and/or low-energy laser or scalp surgery for AGA within 12 months prior to screening;
  12. Have used other medical shampoos or solutions containing ketoconazole or similar ingredients (e.g., Terzolin) that may affect the efficacy evaluation within 1 month prior to screening;
  13. Plan to use any adjuvant or concomitant therapy for the treatment of alopecia throughout the study;
  14. Allergic to the study drug or known to be allergic to ingredients of the study drug;
  15. History of malignant diseases within 5 years prior to screening;
  16. Abnormal and clinically significant findings in physical examination, vital signs, 12-lead ECG, hematology, urinalysis, blood chemistry and thyroid function test at screening, which will affect the efficacy and safety evaluation and study results as judged by the investigator;
  17. Positive for any one or more of antibodies of treponema pallidum antibody, human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen or hepatitis C virus antibody;
  18. Have undergone major surgery within 3 months prior to screening, or plan to undergo major surgery during the study;
  19. Have participated in or being participated in clinical studies of interventional drugs or medical devices within 3 months prior to screening (except for those who participated in non-interventional studies and those who only signed the ICF but did not receive study intervention);
  20. History of drug abuse within 1 year prior to screening, or history of drug use or alcohol dependence within 3 months prior to the study;
  21. Those who, in the opinion of the investigator, have other conditions that may affect compliance or are not suitable for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Assessment of change in Target Area Hair Counts | 24 weeks
  Changes from baseline in non-vellus TAHC (Target Area Hair Counts) in comparison to placebo (Non-vellus TAHC is the number of non-vellus hairs within 1 cm² scalp, which usually ranges from 0 to 300. Larger non-vellus TAHC implies thicker hair. In this study, larger change in non-vellus TAHC means better outcome.)

SECONDARY OUTCOMES:
Assessment of change in Hair Growth Assessment score | 6,12,18 and 24 weeks
  Changes from baseline in HGA (Hair Growth Assessment) score by Principal Investigator and subjects (HGA scale ranged from -3 to 3 and represented decreases from baseline that were substantial, moderate, slight, no change, slight increases, moderate increases, and substantial increases, respectively. HGA improvement was defined as a hair growth assessment score of larger than 0.)

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Dermatology Hospital of Southern Medical University, Guangzhou
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Huashan Hospital, Fudan University, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Suining Central Hospital, Suining
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: No